CLINICAL TRIAL: NCT05744869
Title: School-based Asthma Therapy to Advance Health Equity Among Historically Marginalized Children
Brief Title: SBAT for Health Equity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Michigan State University (Other); Virginia Polytechnic Institute and State University (Other); University at Buffalo (Other)
Responsible Party: Principal Investigator, Jill Halterman, Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00008016
Record Dates: First submitted 2023-01-23; First posted 2023-02-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBAT Implementation (Experimental): For schools randomized to implementing SBAT, the program will include the components already available in comparison (usual care) schools (asthma symptom screening forms, access to telemedicine visits, and protocol for initiating DOT), as well as the following elements that will be facilitated with the support of an implementation team:
  1. telemedicine asthma visits through school with primary care and/or specialist providers to prescribe needed initial medication as well as medication step-ups for DOT
  2. school-based DOT of preventive asthma medications
  3. follow-up telemedicine asthma control assessments
  4. centralized case management support and care coordination
  Interventions: Behavioral: SBAT Implementation
- Usual Care (Active Comparator): During student health services orientation, the SBAT team will recommend school-based DOT for all children with persistent or poorly controlled asthma, and will provide a simple asthma screening survey to assess symptoms and a written protocol for initiating DOT. Telemedicine visits and DOT are available for all children in the school district, but the implementation team will not help to facilitate these components within the usual care schools.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: SBAT Implementation — Implementation of the SBAT Program
  Arms: SBAT Implementation
Behavioral: Usual Care — Usual Care for children with asthma
  Arms: Usual Care

SUMMARY:
The goal of this research trial is to: 1) Solidify a population health SBAT implementation strategy with our longstanding community collaborators, 2) Perform a district-wide hybrid type 3, stepped-wedge, cluster randomized trial, and 3) Assess the supportive resource utilization and essential features of SBAT to extend sustainability and fidelity in a cost-effective manner.

DETAILED DESCRIPTION:
Despite well-established asthma guidelines and availability of effective preventive medications, poor access to guideline-based care is common, especially in historically marginalized communities negatively impacted by social determinants of health (SDOH). There are long-standing inequities in asthma medication use, health care utilization, and outcomes based on race, income, and geography that are rooted in systemic racism and segregation. Many children who should receive daily preventive anti-inflammatory medications do not receive them and follow up care with needed step-ups in asthma treatment does not occur consistently.

Almost 20 years ago, in partnership with the Rochester City School District, an under-resourced urban district with very high poverty rates, the investigators co-developed the paradigm-shifting School-Based Asthma Therapy (SBAT) program to enhance access to guideline-based treatment for children with persistent asthma. SBAT reduces SDOH-related care barriers through the use of: 1) school-based telemedicine visits with primary care providers and asthma specialists facilitating access to asthma assessments for appropriate medication prescription and follow-up, and 2) school-based directly observed therapy (DOT) of preventive asthma medications ensuring access and adherence to these medications. In research studies, SBAT yielded substantial benefit in reducing symptoms and exacerbations, and key stakeholders (caregivers, school district leaders, nurses) express a strong interest in program continuation, since improving asthma outcomes is a top priority for the district and community. Importantly, while this evidence-based program is well accepted in our community and components have been adopted across the country, it has not been implemented broadly in our community nor sustained outside of research trials. SDOH-related barriers have increased over time exacerbating existing health disparities, and children with asthma continue to suffer from morbidity and even mortality. To produce a sustainable public health impact, the investigators must re-imagine school-based asthma care using novel approaches, co-created with our key stakeholders, to define the supports and resources required to extend this evidence-based program's reach and create a resource for national dissemination.

The investigators plan to solidify and test a pioneering SBAT implementation strategy to enhance guideline-based asthma care and reduce disparities. The multilevel SBAT program addresses various SDOH related to healthcare access and quality and social contextual factors that interfere with optimal asthma management. The investigators aim to: 1) Solidify a population health SBAT implementation strategy with our longstanding community collaborators, 2) Perform a district-wide hybrid type 3, stepped-wedge, cluster randomized trial, and 3) Assess the supportive resource utilization and essential features of SBAT to extend sustainability and fidelity in a cost-effective manner.

Upon conclusion, the investigators will have refined and evaluated a stakeholder-driven approach to optimize implementation of SBAT for sustainable improvement in care to ensure health equity for children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma, with persistent symptoms or poor control based on NHLBI criteria
* Age >4 and <12 years
* Attending school in Rochester City School District
* Caregiver >18 years, and is able to understand and speak English or Spanish

Exclusion Criteria:

* Caregiver inability to speak and understand English or Spanish. (*Participants unable to read will be eligible, and all instruments will be given verbally.)
* Having other significant medical conditions, including congenital heart disease, cystic fibrosis, or other chronic lung disease, that could interfere with the assessment of asthma-related measures.
* In foster care or other situations in which consent cannot be obtained from a guardian.

Based on our prior studies, fewer than 10% of subjects are expected to be excluded based on these criteria.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of children on DOT | 3 month follow-up
  The percentage of eligible children in schools initiated on guideline-based DOT at the 3 month follow-up.

IPD SHARING:
Plan to Share IPD: Yes
All raw data produced in the course of the project will be preserved. All de-identified quantitative analysis datasets will be shared once the main study results have been accepted for publication.
  The research data from this project will be deposited within the digital repository of the Inter-university Consortium for Political and Social Research (ICPSR) to ensure that the research community has long-term access to the data, once the main study manuscript has been accepted for publication (or by the end of the grant period; whichever comes first).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available once the results from the main study aims have been accepted for publication or study closure (whichever comes first), and will remain available for 5 years past the grant end date.
Access Criteria: Public-use data files: These files, in which direct and indirect identifiers have been removed to minimize disclosure risk, may be accessed directly through the ICPSR website.
  Restricted-use data files: These files are distributed in those cases when removing potentially identifying information would significantly impair the analytic potential of the data. Users (and their institutions) must request these files from Dr. Halterman and complete a Data Sharing Agreement. The investigator team will review and approve each request.